CLINICAL TRIAL: NCT03820232
Title: Intraoperative Body Core Temperature Monitoring in Patients Undergoing Major Abdominal Surgery: Comparison Between the Oesophageal Probe and the Heated Controlled Servo Sensor
Brief Title: Intraoperative Body Core Temperature Monitoring: Oesophageal Probe vs Heated Controlled Servo Sensor
Acronym: ESOSPOT
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, Principal investigator, Careggi Hospital
Other Study IDs: 11994_spe
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Surgery; Temperature Change, Body
Keywords: Intraoperative, Hypothermia
MeSH Terms: conditions — Body Temperature Changes; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Surgical patients: Patients who were candidates for major or urological surgery under general anaesthesia will be observed. In particular, the core body temperature will be measured with both a single-use oesophageal probe and a SpotOn® heated controlled servo sensor.
  Interventions: Device: temperature monitoring

INTERVENTIONS:
Device: temperature monitoring — In every patient observed in this prospective observational study, body core temperature will be contemporaneously monitored through the oesophageal probe and the heated controlled servo sensor. Both are routinely used for this purpose in clinical practice

SUMMARY:
Monitoring of intraoperative core temperature is essential for patient safety, reducing the risk of perioperative hypothermia. A recently developed measuring system, SpotOn® (3M, St. Paul, MN), measures the core temperature in a non-invasive manner. Its accuracy in patients undergoing general surgery has not been investigated yet. The study was aimed at comparing the accuracy of the SpotOn® in comparison with the oesophageal probe which is considered the current standard in our care units.

DETAILED DESCRIPTION:
Monitoring of intraoperative core temperature is essential for patient safety, reducing the risk of perioperative hypothermia. A recently developed measuring system, SpotOn® (3M, St. Paul, MN), measures the core temperature in a non-invasive manner. Its accuracy in patients undergoing general surgery has not been investigated yet. The study was aimed at comparing the accuracy of the SpotOn® in comparison with the oesophageal probe which is considered the current standard in our care units. In this study, patients who were candidates for major or urological surgery will be considered eligible for enrollment. The core body temperature will be thus measured with both a single-use oesophageal probe and a SpotOn® heated controlled servo sensor.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* patients scheduled for major abdominal surgery
* patients scheduled for general anesthesia
* expected surgery duration longer than 30 minutes

Exclusion Criteria:

* skin infection in the forehead
* upper airway anatomy alterations
* pre-existing oesophageal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were candidates for major or urological surgery were considered eligible to be enrolled. The core body temperature was measured with both a single-use oesophageal probe and a SpotOn® heated controlled servo sensor.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
accuracy of heated controlled servo sensor in monitoring body core temperature compared with oesophageal probe | 1 hour after the induction of general anesthesia
  Difference between temperature measured with heated controlled servo sensor and oesophageal probe

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Villa, Principal Investigator — Azienda Careggi
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morettini E, Turchini F, Tofani L, Villa G, Ricci Z, Romagnoli S. Intraoperative core temperature monitoring: accuracy and precision of zero-heat flux heated controlled servo sensor compared with esophageal temperature during major surgery; the ESOSPOT study. J Clin Monit Comput. 2020 Oct;34(5):1111-1119. doi: 10.1007/s10877-019-00410-z. Epub 2019 Oct 31. PMID 31673946